CLINICAL TRIAL: NCT00005516
Title: Epidemiology of Sleep Disordered Breathing in Children
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5035; R01HL060957 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-03

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes

SUMMARY:
To collect fundamental data regarding the distribution of measures of sleep disordered breathing (SDB) in a pediatric population, prevalence of clinically significant SDB in children, risk factors, and associated co-morbidity.

DETAILED DESCRIPTION:
BACKGROUND:

Developing strategies for recognizing and treating children with Sleep Disordered Breathing (SDB) was not possible in the absence of essential epidemiological data that addressed the distribution of measures of SDB in pediatric populations. The potential public health importance of this was underscored by preliminary data that suggested that risk of SDB was increased in susceptible populations, in particular in African Americans and in children born prematurely.

DESIGN NARRATIVE:

The design was that of a cohort study with a nested case control arm. Sleep disordered breathing was evaluated in 850 children with in-home state-of-the art respiratory monitoring techniques. A number of risk factors were evaluated: sociodemographic characteristics; anthropometry; upper and lower airway size and function (questionnaire, spirometry, and reflectometry); perinatal exposures (from neonatal records); family history; and home environment (passive smoking; sleep patterns, maternal-child stress indices). Behavior, cognitive skills, attention, and health-related quality of life were assessed with standardized instruments to assess co-morbidities (potential SDB outcomes). Analysis of the longitudinal data provided cognitive-developmental trajectories that were evaluated in relationship to SDB. The case-control arm confirmed and extended the findings of the in-home assessments with comprehensive laboratory polysomnography, cephalometry, and objective measures of sleepiness (Multiple Sleep Latency Tests) in three groups of children: definite SDB by home assessment; equivocal SDB; and no SDB. Collection of comprehensive polysomnographic data helped to identify which measures best discriminated symptomatic (e.g., snoring, sleepy) from asymptomatic children.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-07; Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline — Case Western Reserve University

REFERENCES:
- [Background] Monahan KJ, Larkin EK, Rosen CL, Graham G, Redline S. Utility of noninvasive pharyngometry in epidemiologic studies of childhood sleep-disordered breathing. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1499-503. doi: 10.1164/rccm.200111-061OC. PMID 12045123
- [Background] Rosen CL, Palermo TM, Larkin EK, Redline S. Health-related quality of life and sleep-disordered breathing in children. Sleep. 2002 Sep 15;25(6):657-66. PMID 12224844
- [Background] Rosen CL, Larkin EK, Kirchner HL, Emancipator JL, Bivins SF, Surovec SA, Martin RJ, Redline S. Prevalence and risk factors for sleep-disordered breathing in 8- to 11-year-old children: association with race and prematurity. J Pediatr. 2003 Apr;142(4):383-9. doi: 10.1067/mpd.2003.28. PMID 12712055
- [Background] Rosen CL, Storfer-Isser A, Taylor HG, Kirchner HL, Emancipator JL, Redline S. Increased behavioral morbidity in school-aged children with sleep-disordered breathing. Pediatrics. 2004 Dec;114(6):1640-8. doi: 10.1542/peds.2004-0103. PMID 15574628
- [Background] Sulit LG, Storfer-Isser A, Rosen CL, Kirchner HL, Redline S. Associations of obesity, sleep-disordered breathing, and wheezing in children. Am J Respir Crit Care Med. 2005 Mar 15;171(6):659-64. doi: 10.1164/rccm.200403-398OC. Epub 2004 Dec 10. PMID 15591475